CLINICAL TRIAL: NCT07407257
Title: SBRT Tumorjev in Zasevkov v Jetrih in Tumorjev Trebušne Slinavke
Brief Title: SBRT for Liver Tumors, Liver Metastases, and Pancreatic Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OI_SBRT-LIVER-PANCREAS-2019; ERID-KSOPKR-0091/2019 (Other: Ethics Committee, Institute of Oncology Ljubljana)
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Liver Neoplasms; Liver Metastases; Pancreatic Neoplasms
Keywords: SBRT; stereotactic body radiotherapy; liver tumor; pancreatic tumor
MeSH Terms: conditions — Liver Neoplasms; Pancreatic Neoplasms; Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT Treatment (Experimental): Patients with liver tumors, liver metastases, or pancreatic tumors treated with stereotactic body radiotherapy (SBRT) according to the institutional protocol.
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy (SBRT) — Stereotactic body radiotherapy (SBRT) delivered according to the institutional protocol for treatment of liver tumors, liver metastases, and pancreatic tumors, with high-dose hypofractionated radiation and image-guided radiotherapy techniques.

SUMMARY:
This prospective observational study evaluates the safety and effectiveness of stereotactic body radiotherapy (SBRT) for liver tumors, liver metastases, and pancreatic tumors. The study focuses on systematic monitoring and optimization of the SBRT treatment process, including adherence to the implemented protocol, with the aim of simplifying methods while maintaining treatment safety.

DETAILED DESCRIPTION:
Stereotactic body radiotherapy (SBRT) is an advanced radiotherapy technique that enables delivery of high radiation doses to tumors with high precision while limiting exposure of surrounding healthy tissues. This study prospectively follows patients treated with SBRT for primary liver tumors, liver metastases, and pancreatic tumors at the Institute of Oncology Ljubljana.

The primary aim is to monitor and optimize all steps of the SBRT workflow, including protocol adherence, in order to ensure safe implementation and to evaluate treatment outcomes. The study also aims to assess whether the established SBRT protocol can be simplified without compromising patient safety.

Treatment safety and effectiveness outcomes will be evaluated during follow-up, and the collected data will be used to support further refinement of SBRT procedures for upper gastrointestinal tumors

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years

Patients with liver tumors, liver metastases, or pancreatic tumors eligible for stereotactic body radiotherapy (SBRT)

Planned treatment with SBRT according to institutional protocol

Ability to comply with treatment and follow-up procedures

Signed informed consent

Exclusion Criteria:

Contraindications for SBRT according to institutional radiotherapy protocol

Prior radiotherapy that prevents safe SBRT delivery to the target region

Severe uncontrolled comorbidities preventing safe SBRT treatment

Pregnancy

Inability to provide informed consent or comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Treatment Safety (Radiotherapy-Related Toxicity) | From start of SBRT up to 12 months after treatment
  Assessment of acute and late treatment-related toxicity after stereotactic body radiotherapy (SBRT) for liver tumors, liver metastases, and pancreatic tumors, evaluated according to standard toxicity criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No